CLINICAL TRIAL: NCT01267812
Title: A Phase II Study of Weekly Maintenance Bortezomib and Rituximab in Mantle Cell Lymphoma Post Autologous Hematopoietic Cell Transplantation
Brief Title: Bortezomib and Rituximab in Treating Patients With Mantle Cell Lymphoma Who Have Previously Undergone Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10137; NCI-2010-02343 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-12-27; First posted 2010-12-29 (Estimated); Results first posted 2022-02-04 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Contiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Recurrent Mantle Cell Lymphoma; Stage I Mantle Cell Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bortezomib; Rituximab; Immunohistochemistry; Gene Expression Profiling; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (bortezomib and rituximab) (Experimental): Doses of bortezomib given is 1.3 mg/m2 weekly x 4 weeks given every 3 month x 8 cycles. Doses of RITUXAN given is 375 mg/m2 give weekly x 4 weeks given every 6 month for 4 cycles.
  Interventions: Drug: bortezomib; Biological: rituximab; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: RNA analysis; Genetic: gene expression analysis; Genetic: DNA analysis; Other: pharmacological study; Other: pharmacogenomic studies; Other: Questionnaire Administration

INTERVENTIONS:
Drug: bortezomib — Given SC or IV
  Other Names: LDP 341; MLN341; VELCADE
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Other: laboratory biomarker analysis — Correlative studies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: RNA analysis — Correlative studies
Genetic: gene expression analysis — Correlative studies
Genetic: DNA analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: pharmacogenomic studies — Correlative studies
  Other Names: Pharmacogenomic Study
Other: Questionnaire Administration
  Other Names: Ancillary Studies

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving bortezomib together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib and rituximab together works in treating patients with mantle cell lymphoma who have previously undergone stem cell transplantation

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the two year disease free survival in mantle cell lymphoma (MCL) patients treated with bortezomib + rituximab after hematopoietic stem cell transplantation (HSCT).

SECONDARY OBJECTIVES:

I. To evaluate the toxicity profile, safety, overall survival, time to treatment failure, remission duration, and biological markers of mantle cell lymphoma patients treated with bortezomib + rituximab after autologous hematopoietic stem cell transplantation.

OUTLINE: Patients receive bortezomib subcutaneously (SC) or intravenously (IV) over 3-5 seconds and rituximab IV on days 1, 8, 15, and 22. Treatment with bortezomib repeats every 3 months for up to 8 courses and treatment with rituximab repeats every 6 months for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological documented or cytological confirmed mantle cell lymphoma; cyclin D1 must be present as evidenced by either fluorescence in situ hybridization (FISH) or immunohistochemical staining
* Patients must have undergone autologous hematopoietic stem cell transplantation (AHCT) and achieved engraftment by day (D)60-180 as evidenced by absolute neutrophil count (ANC) > 1000/mcL and platelets (Plt) > 75,000/mcL
* Patients must be in complete remission at D60-180 after AHCT as evidenced by computed tomography (CT) scan of the neck/chest/abdomen (abd)/pelvis or CT/positron emission tomography (PET) scans
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* Male subject agrees to use an acceptable method for contraception for the duration of the study
* Life expectancy of greater than 3 months
* Karnofsky > 60%
* ANC > 1000/mcL
* Plts > 75,000/mcL
* Total bilirubin within normal institutional limits, patients with elevation of unconjugated bilirubin alone, as in Gilbert's disease, are eligible
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5 x institutional upper limit of normal
* Creatinine up to and including 2 mg/dL

Exclusion Criteria:

* Patient has >= grade 2 peripheral neuropathy within 14 days before enrollment and at D60-180 after AHCT; patients who had >= grade 2 peripheral neuropathy within 14 days before enrollment but resolves to grade 1 or lower peripheral neuropathy at D60-D180 after AHCT can be enrolled at this time
* Patient has > 1.5 x upper limit of normal (ULN) total bilirubin unless history of Gilbert's syndrome
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiographic (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Patient has hypersensitivity to bortezomib, boron or mannitol
* Female subject is pregnant or breast-feeding; confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Patient has received other investigational drugs with 14 days before treatment of treatment with bortezomib + rituximab
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Patients with other active malignancies (no evidence of other cancer or life expectancy greater than 5 years) are ineligible for this study
* Human immunodeficiency virus (HIV) positive patients or hepatitis B or C positive patients
* Patients with active central nervous system (CNS) disease or history of brain metastases (mets) are excluded from study
* Prior exposure to either bortezomib or rituximab is not an exclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-10-03 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mei, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Chen RW, Palmer JM, Tomassetti S, Popplewell LL, Alluin J, Chomchan P, Nademanee AP, Siddiqi T, Tsai NC, Chen L, Zuo F, Abary R, Cai JL, Herrera AF, Rossi JJ, Rosen ST, Forman SJ, Kwak LW, Holmberg LA. Multi-center phase II trial of bortezomib and rituximab maintenance combination therapy in patients with mantle cell lymphoma after consolidative autologous stem cell transplantation. J Hematol Oncol. 2018 Jun 28;11(1):87. doi: 10.1186/s13045-018-0631-3. PMID 29954415

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Bortezomib and Rituximab): Doses of bortezomib given is 1.3 mg/m^2 weekly x 4 weeks given every 3 month x 8 cycles. Doses of RITUXAN given is 375 mg/m^2 give weekly x 4 weeks given every 6 month for 4 cycles.
  bortezomib: Given SC or IV
  rituximab: Given IV
  laboratory biomarker analysis: Correlative studies
  immunohistochemistry staining method: Correlative studies
  RNA analysis: Correlative studies
  gene expression analysis: Correlative studies
  DNA analysis: Correlative studies
  pharmacological study: Correlative studies
  pharmacogenomic studies: Correlative studies
  Questionnaire Administration
Period: Overall Study
Arm/Group | Treatment (Bortezomib and Rituximab)
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Bortezomib and Rituximab): Doses of bortezomib given is 1.3 mg/m2 weekly x 4 weeks given every 3 month x 8 cycles. Doses of RITUXAN given is 375 mg/m2 give weekly x 4 weeks given every 6 month for 4 cycles.
  bortezomib: Given SC or IV
  rituximab: Given IV
  laboratory biomarker analysis: Correlative studies
  immunohistochemistry staining method: Correlative studies
  RNA analysis: Correlative studies
  gene expression analysis: Correlative studies
  DNA analysis: Correlative studies
  pharmacological study: Correlative studies
  pharmacogenomic studies: Correlative studies
  Questionnaire Administration
Arm/Group | Treatment (Bortezomib and Rituximab)
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 59 [45 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Two-year Disease-free Survival
Description: Assessed by Kaplan-Meier survival analysis. 95% confidence intervals will be calculated using Greenwood's formula.
Time Frame: Participants were followed up to 5 years after initial treatment and Kaplan-Meier survival analysis was used to generate the two-year disease-free survival estimate presented.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment (Bortezomib and Rituximab): Doses of bortezomib given is 1.3 mg/m^2 weekly x 4 weeks given every 3 month x 8 cycles. Doses of RITUXAN given is 375 mg/m^2 give weekly x 4 weeks given every 6 month for 4 cycles.
  bortezomib: Given SC or IV rituximab: Given IV
Arm/Group | Treatment (Bortezomib and Rituximab)
Number analyzed (Participants) | 23
percentage of participants | 90 [66 to 97]

2. Secondary Outcome: Two-year Overall Survival
Description: Assessed by Kaplan-Meier survival analysis. 95% confidence intervals will be calculated using Greenwood's formula.
Time Frame: Participants were followed up to 5 years after initial treatment and Kaplan-Meier survival analysis was used to generate the two-year overall survival estimate presented.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Bortezomib and Rituximab)
Number analyzed (Participants) | 23
percentage of participants | 95 [68 to 99]

3. Secondary Outcome: Grade 3 or 4 Toxicities of Bortezomib and Rituximab Treatment
Description: Observed toxicities will be summarized in terms of type, severity (graded by NCI CTCAE version 4.0) and attribution.
Time Frame: Participants were followed up to 5 years after initial treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bortezomib and Rituximab)
Number analyzed (Participants) | 23
Participants
  Neutropenia | 17
  Lymphopenia | 8
  Pneumonia | 2
  Anemia | 2
  Lung infection | 2
  Skin infection | 1
  Wound infection | 1
  Hypertension | 1
  Thrombocytopenia | 1

ADVERSE EVENTS:
Time Frame: Up to five years after initial treatment
Arm/Group | Treatment (Bortezomib and Rituximab)
All-Cause Mortality (participants affected / at risk) | 3/23
Serious Adverse Events (participants affected / at risk) | 7/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bortezomib and Rituximab) (N=23)
Neutrophil Count Decreased (Investigations) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Fever (General disorders) | 2 (2)
Myelodysplastic Syndrome (Blood and lymphatic system disorders) | 1 (1)
Human Metapneumovirus Infection (Infections and infestations) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bortezomib and Rituximab) (N=23)
Anemia (Blood and lymphatic system disorders) | 15 (46)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 6 (7)
Tinnitus (Ear and labyrinth disorders) | 5 (6)
Endocrine disorders - Other, specify (Endocrine disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 3 (4)
Watering eyes (Eye disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Bloating (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 11 (16)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (9)
Vomiting (Gastrointestinal disorders) | 3 (4)
Chills (General disorders) | 8 (9)
Edema limbs (General disorders) | 4 (5)
Fatigue (General disorders) | 21 (38)
Fever (General disorders) | 9 (13)
Flu like symptoms (General disorders) | 2 (2)
Gait disturbance (General disorders) | 3 (5)
Injection site reaction (General disorders) | 8 (9)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 5 (5)
Allergic reaction (Immune system disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 2 (3)
Eye infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 3 (4)
Skin infection (Infections and infestations) | 3 (3)
Upper respiratory infection (Infections and infestations) | 7 (12)
Wound infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 8 (23)
Alkaline phosphatase increased (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 9 (19)
Blood bilirubin increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 6 (17)
Investigations - Other, specify (Investigations) | 5 (37)
Lymphocyte count decreased (Investigations) | 12 (84)
Neutrophil count decreased (Investigations) | 20 (67)
Platelet count decreased (Investigations) | 17 (59)
Weight gain (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 20 (89)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 4 (5)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (10)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 6 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (8)
Obesity (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (5)
Paresthesia (Nervous system disorders) | 6 (6)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 13 (26)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (6)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (19)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 (6)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 17 (43)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT01267812/Prot_SAP_000.pdf